CLINICAL TRIAL: NCT01280799
Title: Acceptance Based Separated Family Treatment for Adolescents With Anorexia Nervosa
Brief Title: Family Treatment for Adolescents With Anorexia Nervosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Towson University (Other)
Collaborators: University of the Sciences in Philadelphia (Other); Duke University (Other)
Responsible Party: Principal Investigator, C. Alix Timko, Assistant Professor, Towson University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH08597
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Anorexia Nervosa; Subthreshold Anorexia Nervosa; Eating Disorder Not Otherwise Specified, Primarily Restriction
Keywords: Anorexia Nervosa; Adolescents; Family Treatment; Eating Disorder; Acceptance and Commitment Therapy
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Treatment (Experimental)
  Interventions: Behavioral: Acceptance-based separated family treatment

INTERVENTIONS:
Behavioral: Acceptance-based separated family treatment — Family treatment that combines Acceptance and Commitment Therapy (ACT) for the adolescent with Parent Skills Training for caregivers. The treatment package is designed to increase willingness to experience difficult thoughts, feelings, and bodily sensations in order to engage in effective behavior. To facilitate this, caregivers are provided with psychoeducation on eating disorders and skills in behavior management, self-regulation, and emotion regulation.

SUMMARY:
This treatment development study seeks to investigate the most effective way to treat an adolescent's eating disorder and how best to involve the parents or caregivers in this process.

Typically, parents and their child are seen together in therapy. However, this can sometimes be difficult for both the parents and the adolescent. Both parents and adolescents have different concerns and are struggling with different aspects of the eating disorder. Therefore, the treatment in this study involves the parents in treatment, but the majority of therapy sessions are conducted with the parent(s) and adolescent separately.

Participants meet with a therapist for 20 sessions over the course of 24 weeks. For the first 16 weeks parents and the adolescent meet individually with the therapist. For the last 8 weeks families meet with the therapist every other week. These last four sessions are conjoint - that is, adolescents and parents will meet with the therapist together. This is to help parents and adolescents come together as a family to continue to aid the adolescent in the treatment of his/her eating disorder.

The investigators hypothesize that adolescents who receive this treatment will demonstrate improvement in eating disorder symptoms and body-mass index and that caregivers who participate will demonstrate decreased distress and caregiver burden. Furthermore, the investigators hypothesize that increases in psychological acceptance will be seen for both adolescents and caregivers post-treatment, and that treatment will be viewed as both credible and acceptable to both caregiver and adolescent.

DETAILED DESCRIPTION:
The purpose of this study is to develop and gather preliminary data on an acceptance-based behavioral treatment for adolescents with anorexia nervosa (AN) that is delivered in a separated family format. The treatment will combine a parent's skills curriculum that has demonstrated preliminary effectiveness in the treatment of AN, with a novel adolescent component based on Acceptance and Commitment Therapy (ACT). ACT has been found to be useful in the treatment of an array of psychological difficulties, and may be particularly well-suited for the cognitive and behavioral avoidance and rigidity that characterizes individuals with AN and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent is between 12-18 years of age and living in home with caregivers
* Parent or primary caregiver willing to attend therapy sessions
* Adolescent meets diagnostic criteria of anorexia nervosa (either restricting or binge/purge subtype) or subthreshold AN (relaxation of weight criterion to 90% of ideal body weight as determined by weight history and CDC growth curves) or eating disorder not otherwise specified (with restricting as the primary symptom) according to the DSM-IV TR
* Adolescent is appropriate for outpatient care and receives medical clearance from a primary care physician

Exclusion Criteria:

* Caregiver or adolescent with a co-morbid diagnosis of psychotic disorder, bi-polar disorder, or substance dependence
* Caregiver or adolescent with diagnosis of mental retardation or a pervasive developmental disorder
* Adolescent with a diagnosis of eating disorder not otherwise specified with the primary symptoms of bingeing and purging, binging without compensatory behaviors or spitting food or with restricting patterns but a BMI greater than 90% ideal weight (as determined by weight history and CDC growth curves)
* Adolescent with extreme malnutrition or other medical complications/ diagnoses that require a higher level of care
* Acute suicide risk

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI | 9 months (6 months active treatment, 3 months follow-up)

SECONDARY OUTCOMES:
Eating Disorder Examination (16.0D) | 9 months (6 months of treatment and 3 month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Alix Timko, PhD, Principal Investigator — Towson University/University of the Sciences
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of the Sciences, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Timko CA, Zucker NL, Herbert JD, Rodriguez D, Merwin RM. An open trial of Acceptance-based Separated Family Treatment (ASFT) for adolescents with anorexia nervosa. Behav Res Ther. 2015 Jun;69:63-74. doi: 10.1016/j.brat.2015.03.011. Epub 2015 Mar 28. PMID 25898341